CLINICAL TRIAL: NCT01919879
Title: A Multicentric Randomized Phase II Trial Evaluating Dual Targeting of EGFR Using the Combination of Cetuximab and Afatinib Versus Cetuximab Alone in Patients With Chemotherapy Refractory wtKRAS Metastatic Colorectal Cancer
Brief Title: Dual Targeting of EGFR With Cetuximab and Afatinib to Treat Refractory wtKRAS Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UCGI 25
Record Dates: First submitted 2013-03-01; First posted 2013-08-09 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Chemotherapy refractory; wtKRAS metastatic colorectal cancer; cross over
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Cetuximab + Afatinib (Experimental): Afatinib 40 mg daily Cetuximab 500 mg/m2 every 2 weeks until progression
  Interventions: Drug: Cetuximab + Afatinib
- Arm B : Cetuximab alone (Active Comparator): Cetuximab 500mg/m2 every 2 weeks until progression After progression: Cetuximab 500mg/m2 + Afatinib 40 mg per day until progression
  Interventions: Drug: Cetuximab + Afatinib; Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab + Afatinib — Afatinib taken orally, cetuximab administered intravenously
  Other Names: Erbitux
Drug: Cetuximab — Cetuximab administered intravenously
  Other Names: Erbitux
  Arms: Arm B : Cetuximab alone

SUMMARY:
This is a multicentric, phase II and open label study.75 patients are expected to be randomized in 35 centers. The main objective is to assess the efficacy and safety of Afatinib -cetuximab combo versus cetuximab alone in treatment of patients with refractory wtKRAS metastatic colorectal cancer.

DETAILED DESCRIPTION:
Patients who will sign the inform consent will be enrolled into one of two groups. Group A will receive Afatinib ( 40mg per day) and Cetuximab (500mg/m2)every two weeks until progression. Group B will receive Cetuximab (500mg/m2) alone every two weeks until progression and after progression,patients from group B will receive afatinib (group A treatment) until progression. The criteria for evaluation will be tumor response and progression documented by CT scan and according to RECIST criteria version 1.1.

Patient will also sign a inform consent before participating in biological study. The aim of this translational study is to collect tumor and blood sample in order to determine, the biological factors which are predictive of the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic colorectal cancer expressing the wtKRAS status
2. No previous EGFR targeted therapy.
3. Must have failed a prior regimen containing irinotecan for metastatic disease and a prior regimen containing oxaliplatin for metastatic disease
4. Must have previously received a thymidylate synthase inhibitor (eg, fluorouracil, capecitabine, raltitrexed, or fluorouracil-uracil) at any point for treatment of colorectal cancer (CRC)
5. Life expectancy of at least 3 months.
6. Patient with ECOG ≤ 1
7. Patients aged ≥ 18.
8. Patient with measurable lesions according to RECIST criteria (version 1.1) with spiral CT scan and defined as ≥ 10 mm in longest diameter and 2X the slice thickness for extra nodal lesions and/or > 15 mm in short axis diameter for nodal lesions
9. Patient able to receive adequate oral nutrition of ≥ 1500 calories per day and free of significant nausea and vomiting
10. Patient with adequate organ function:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Haemoglobin ≥ 9 g/dL
    * Platelets (PTL) ≥ 100 x 109/L
    * AST/ALT ≤ 3 x ULN (≤ 5 x ULN in case of liver metastases)
    * GammaGT < 3 x ULN (< 5 x ULN in case of liver involvement)
    * Bilirubin ≤ 1.5 x ULN
    * Creatinine clearance ≥ 50 mL/min (Cockcroft and Gault formula)
11. Adequate contraception if applicable.
12. Ability to take oral medication in the opinion of the investigator
13. Patient able and willing to comply with study procedures as per protocol
14. Patient able to understand and willing to sign and date the written voluntary informed consent form at screening visit prior to any protocol-specific procedures
15. Patient affiliated to a social security regimen

Exclusion Criteria:

1. Previous EGFR targeted therapy.
2. Mutant KRAS status
3. Prior severe reaction to a monoclonal antibody
4. No heart failure or coronary heart disease symptoms Clinically relevant cardiovascular abnormalities, as judged by the investigator, such as, but not limited to, uncontrolled hypertension, congestive heart failure NYHA classification > III, unstable angina, myocardial infarction within six months prior to randomisation, or poorly controlled arrhythmia
5. Cardiac left ventricular dysfunction with resting ejection fraction of less than institutional lower limit of normal (if no lower limit of normal is defined in the institution, the lower limit is 50%)
6. Symptomatic brain metastases requiring treatment
7. Major surgery within 28 days or minor surgery within 14 days of the start of the study treatment
8. Radiotherapy less than two weeks prior to the start of the study treatment
9. Systemic chemotherapy, hormonal therapy, immunotherapy ≤ 21 days before study treatment
10. No major comorbidity that may preclude the delivery of treatment or active infection (HIV or chronic hepatitis B or C) or uncontrolled diabetes.
11. Concomitant occurrence of another cancer, or history of cancer within the past five years except in situ carcinoma of the cervix treated or basal cell carcinoma or squamous cell carcinoma.
12. Known pre-existing interstitial lung disease
13. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease, malabsorption, or CTCAE grade >2 diarrhea of any etiology
14. Pregnant woman or lactating woman.
15. Persons deprived of liberty or under guardianship.
16. Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
17. Previous history of keratitis, ulcerative keratitis or severe dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Non progression rate at 6 months | 6 months
  The progression rate is defined as percentage of patients without progression at 6 months after observation of all patients at 6 months

SECONDARY OUTCOMES:
Overall response rate (OR) | 6 months
  Overall response rate is defined as percentage of subjects with a confirmed complete or partial response as per RECIST V1.1 criteria
Progression free survival | until progression or death, expected average approximately 4 months
  It is define as the time of from randomization to date of first documented progression or any cause of death
Overall and specific survival | until death, on average approximately 14 months
  Overall and specific survival is defined from time of randomization to the date of documented death
Quality of life | During treatment, on average approximately 4 months
  EORTC QLQ-C30 and QLQ-CR29 are questionnaires developed to assess the quality of life of cancer patients
Tolerance of the treatment | until progression, expected approximately 4 months
  Safety of the study treatment will be assessed on occurrence of Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Helene SENELLART, Dr, Principal Investigator — Centre René Gauducheau- Nantes Saint herbelain; Evelyne BOUCHER, Dr, Principal Investigator — Centre Eugène Marquis-Rennes; Eric FRANCOIS, Dr, Principal Investigator — Centre Antoine Lacassagne, Nice; Emmanuelle SAMALIN SCALZI, Dr, Principal Investigator — Centre Val d'Aurel-Paul Lamarque-Montpellier; Meher BEN ABDELGHANI, Dr, Principal Investigator — Centre Paul Strauss-Strasbourg; Antoine ADENIS, Pr, Principal Investigator — Centre Oscar Lambret_Lille; Christelle DE LA FOUCHARDIERE, Dr, Principal Investigator — Centre Léon Bérard, Lyon; François GHIRENGHELLI, Dr, Principal Investigator — Centre Georges Leclerc-Dijon; Olivier DUBROEUCQ, Dr, Principal Investigator — Centre Jean Godinot-Reims; Emmanuelle MITRY, Dr, Principal Investigator — Hopital Rene Huguenin_Intitut Curie_Paris; Christophe BORG, Pr, Principal Investigator — Hôpital Jean Minjoz-Besaçon; Yves BOUCARN, Dr, Principal Investigator — Institut Bergonié Bordeaux; Christophe BORG, Pr, Principal Investigator — Centre Hospitalier de Belfort-Montbelliard; Marion CHAUVENET, Dr, Principal Investigator — Centre Hospitalier Lyon Sud-Pierre Benite
Locations (1):
- Institute de Cancérologie de la Loire, Nantes, France